CLINICAL TRIAL: NCT07005726
Title: BCG2-DTP3: Providing BCG Revaccination With the Third Dose of Diphtheria-tetanus-pertussis Vaccine to Improve Female Survival in Africa
Brief Title: BCG Revaccination With the Third Dose of Diphtheria-tetanus-pertussis Vaccine and Infant Mortality in Africa
Acronym: BCG2-DTP3
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: University of Southern Denmark (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 003/CNES/INASA/2025
Record Dates: First submitted 2025-05-05; First posted 2025-06-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Infant Morbidity; Infant Mortality; Non-Specific Effects of Vaccines; BCG
Keywords: Non-specific-effects of vaccines; BCG; DTP; Infant mortality; Guinea-Bissau; Infant morbidity; Female survival; BCG revaccination
MeSH Terms: conditions — Infant Death | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All follow-up will be masked as the intervention is not marked on the child's vaccination card.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG2+DTP3 (Experimental): Infants aged 14-24 weeks will receive a second dose of BCG with the third dose of DTP.
  Interventions: Biological: BCG Vaccine
- DTP3 (No Intervention): Infants aged 14-24 weeks will as-per-usual receive a third dose of DTP.

INTERVENTIONS:
Biological: BCG Vaccine — The WHO-prequalified BCG-Japan or BCG-Denmark
  Arms: BCG2+DTP3

SUMMARY:
Studies in low-income countries show that vaccines can have important non-specific effects on other infections. Live BCG vaccine can train the immune system and reduce susceptibility to unrelated infections. In contrast, non-live diphtheria-tetanus-pertussis-containing (DTP) vaccine enhances susceptibility in females: DTP vs no DTP is associated with 2-fold higher mortality, and in DTP-vaccinated children, females have higher mortality than males. These effects are seen as long as a vaccine is the most recent vaccine. WHO recommends BCG at birth followed by three DTP vaccines. A metaanalysis based on observational studies has shown that co-administration of BCG+DTP is associated with lower mortality than BCG followed by DTP.

The investigators will implement a randomised trial in urban Guinea-Bissau, including 6000 children, to test the hypothesis that an extra dose of BCG given with DTP3 (BCG2+DTP3 vs. DTP3) can:

* reduce death and hospital admissions by 25%
* reduce the F/M severe morbidity hazard ratio

DETAILED DESCRIPTION:
Background:

Since the 1970s, the basic vaccination schedule in low-income countries has sequenced BCG and DTP, so that BCG was provided at birth and diphtheria-tetanus-pertussis vaccine (DTP, now in a version with H. influenza vaccine and hepatitis B, 'pentavalent vaccine') in 3 doses at 6,10, and 14 weeks, followed by measles vaccine (MV) at 9 months of age.

WHO recommends DTP-after-BCG but a meta-analysis of observational studies has shown that co-administration of BCG+DTP is associated with 43% (27-54%) lower mortality than DTP after BCG (Higgins et al, BMJ 2016).

The idea that vaccines can change morbidity and mortality in ways not explained by prevention of the vaccine-targeted infection is gaining increasing recognition. Major examples of beneficial NSEs include that the live BCG vaccine reduces non-tuberculosis infections. In contrast, the non-live DTP vaccine is associated with increased susceptibility to non-DTP infections and higher female mortality.

When WHO reviewed the NSEs of vaccines, the DTP vaccine was associated with a 38% (-8-108%) increase in mortality, but providing BCG-with-DTP was associated with 48% (30-66%) lower mortality than the usual schedule of BCG-then-DTP.

Based on this evidence, the investigators propose an randomised controlled trial (RCT) to test whether co-administration of a second dose of BCG (BCG2) with the third dose of DTP (DTP3) reduces the severe morbidity rate and the F/M HR.

Hypotheses:

* BCG2+DTP3 vs. DTP3 reduces severe morbidity, i.e. non-accidental deaths and hospital admissions, by 25% until MV is given.
* BCG2+DTP3 vs. DTP3 reduces the F/M severe morbidity hazard ratio until MV is given.

Methods:

The RCT will be nested within the Bandim Health Project (BHP) Health and Demographic Surveillance System (HDSS) study area. The RCT will be conducted in the urban areas of the BHP HDSS, which follows approximately 100,000 inhabitants (www.bandim.org). The BHP registers pregnancies, births, and follow young children until 3 years of age. During home visits, data is collected regarding infections, hospitalisations, vaccinations, breastfeeding, growth, and survival. At the first contact, BHP assistants provide a vaccination card for the child, which serves as an ID card during subsequent health system contacts. At the home visits, mothers are encouraged to bring their children for vaccination. All vaccinations and consultations at the three health centres in the study area are documented. Furthermore, BHP registers deliveries and paediatric consultations and admissions at the Simão Mendes national hospital.

When the child is approaching 14 weeks of age, written (Portuguese) and verbal (Creole Portuguese) information will be provided during a home visit. Children, who are not seriously ill and whose parents are willing to take part, will be invited to the health centre for enrolment (see exclusion/inclusion criteria below).

At the centre, participants will be asked to obtain oral and written consent. It will be explained that the Ministry of Health does not routinely recommend BCG2. However, studies from several countries suggest that BCG can improve health. Therefore, it will be examined whether the addition of BCG2 contributes to better child health. Those who wish to take part in the study are asked to sign consent forms (or in case of illiteracy provide thumb print on consent forms).

The child's vaccination card will be transcribed, and the child will be examined by a clinician. Both mother and child will be examined for BCG-scars. Finally, the children will be randomised to BCG or no intervention (1:1 in blocks, stratified by sex, to BCG or no intervention with DTP3 using REDCap).

The investigators will not record BCG2/no intervention on the child's vaccination card, and all field assistants and hospital workers collecting outcome data will be unaware of the child's allocation. The mothers/guardians of participating children will know whether the child received BCG or No Intervention.

Enrolled children will be called every 2 months to assess vital status, hospitalizations and consultations. In case telephone contact is not achieved, a home visit will be conducted. At 9 months of age all children will be visited at home and invited to the health centre for clinical assessment.

Deaths are detected at the regular contacts. Within 3 months after a death, the family will be interviewed to conduct a verbal autopsy (VA). The cause of death will be based on the physician diagnosis for in-hospital deaths or the VA-history for children that died elsewhere. Based on this information, deaths will be classified as accidental or non-accidental.

Most admissions occur at the national paediatric ward and will be registered there by the BHP staff. At the regular contacts, the mother will be asked whether the child has been hospitalised. A questionnaire is completed for each admission to obtain timing, symptoms, duration, and place of admission. Admissions will be counted as non-accidental if the paediatric ward data indicates that it was not caused by an accident.

With a mortality risk of 1.5% and a hospitalisation risk of 7.5% between 14 weeks and 9 months, the study can detect a 25% reduction in deaths and hospitalisations with 4700 participants (power 80%; significance 5%). With a 9% risk of the composite outcome, there will be have considerable power to detect minor changes in the F/M severe morbidity ratio. Over 4-5 years of enrolment, the plan is to recruit 6000 children, allowing for loss to follow-up and potential interference from national campaigns.

Statistical analyses:

Cox regression models will be used to compare severe morbidity for BCG2+DTP3 versus controls (No intervention+DTP3). Children are followed from enrolment until death, migration, measles vaccination, age 12 months, or end of study. Potential effect modifiers will be investigated. Since vaccines interact, follow-up in the main analysis will be censored at vaccination campaigns and this could reduce the power of the study. However, OPV is the only vaccine used in campaigns in this age group and these campaigns are now rare.

All comparisons of BCG2+DTP3 vs No intervention+DTP3 will be analysed separately by sex. Potential effect modifiers besides sex include season, vaccination campaigns, BCG status, and BCG scar status of mother and child prior to enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Children, who are between 14 weeks and 24 weeks of age,
* Received DTP2 at least 4 weeks earlier and who are due to receive DTP3.

Exclusion Criteria:

* Children, who are ill and require hospitalization.
* Children with severe malformations
* Children, who had suppurative lymphadenitis after BCG1 (extremely rare)

Ages: 14 Weeks to 24 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6000 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Non-accidental servere morbidity | Baseline to the age of measles vaccine (scheduled at 9 months, to be received by latest by 12 months. Children will be censored upon migration or death.
  Composite outcome of death and admissions. Obtained via active follow-up of participants by phone calls, home visits and at the hospital.
  Cox regression models will be used to compare severe morbidity for BCG2+DTP3 versus controls (DTP3).
  The comparison of BCG2+DTP3 vs DTP3 will also be analysed separately by sex

SECONDARY OUTCOMES:
Female/Male servere morbidity ratio | Baseline to the age of measles vaccine (scheduled at 9 months, to be received by latest by 12 months. Children will be censored upon migration or death.
  Composite outcome of death and admissions. Obtained via active follow-up of participants by phone calls, home visits and at the hospital.
  Cox regression models specified by sex will be used to compare severe morbidity for BCG2+DTP3 versus controls (DTP3).
Non-accidental mortality | Baseline to the age of measles vaccine (scheduled at 9 months, to be received by latest by 12 months. Children will be censored upon migration or death.
  Information obtained via active follow-up of participants by phone calls, home visits and at the hospital.
  Cox regression models will be used to compare mortality for BCG2+DTP3 versus controls (DTP3).
  The comparison of BCG2+DTP3 vs DTP3 will also be analysed separately by sex
Non-accidental morbidity | Baseline to the age of measles vaccine (scheduled at 9 months, to be received by latest by 12 months. Children will be censored upon migration or death.
  Information obtained via active follow-up of participants by phone calls, home visits and at the hospital. Cox regression models will be used to compare hospital admissions for BCG2+DTP3 versus controls (DTP3).
  The comparison of BCG2+DTP3 vs DTP3 will also be analysed separately by sex
Cause-specific deaths | Baseline to the age of measles vaccine (scheduled at 9 months, to be received by latest by 12 months. Children will be censored upon migration or death.
  Information obtained via active follow-up of participants by phone calls, home visits and at the hospital. Cox regression models will be used to compare cause-specific mortality for BCG2+DTP3 versus controls (DTP3).
  The comparison of BCG2+DTP3 vs DTP3 will also be analysed separately by sex.
Cause-specific admissions | Baseline to the age of measles vaccine (scheduled at 9 months, to be received by latest by 12 months. Children will be censored upon migration or death.
  Information obtained via active follow-up of participants by phone calls, home visits and at the hospital. Cox regression models will be used to compare cause-specific hospital admissions for BCG2+DTP3 versus controls (DTP3).
  The comparison of BCG2+DTP3 vs DTP3 will also be analysed separately by sex.
Consultations | Baseline to the age of measles vaccine (scheduled at 9 months, to be received by latest by 12 months. Children will be censored upon migration or death.
  Information obtained via active follow-up of participants by phone calls, home visits and at the hospital. Cox regression models will be used to compare out-patient consultations for BCG2+DTP3 versus controls (DTP3).
  The comparison of BCG2+DTP3 vs DTP3 will also be analysed separately by sex.
Adverse reactions in a subset of 800 participants | From baseline to baseline+6 months
  A morbidity study of the first 800 children will be conducted, using weekly (month 1) and monthly (months 2-6) morbidity interviews by phone in addition to data on admissions at the national hospital to assess potential adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Stabell Benn, MD, PhD, DMSc, Principal Investigator — Bandim Health Project and Danish Institute for Advanced Science, University of Southern Denmark
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No
Deidentified participant data with a data dictionary can be shared after approval of a data-sharing proposal sent to Professor Christine Stabell Benn (cbenn@health.sdu.dk) and approval by the the Guinea-Bissau Ethical Committee for Health Research

REFERENCES:
- [Background] Aaby P, Ravn H, Benn CS. The WHO Review of the Possible Nonspecific Effects of Diphtheria-Tetanus-Pertussis Vaccine. Pediatr Infect Dis J. 2016 Nov;35(11):1247-1257. doi: 10.1097/INF.0000000000001269. PMID 27753772
- [Background] Aaby P, Nielsen J, Benn CS, Trape JF. Sex-differential and non-specific effects of routine vaccinations in a rural area with low vaccination coverage: an observational study from Senegal. Trans R Soc Trop Med Hyg. 2015 Jan;109(1):77-84. doi: 10.1093/trstmh/tru186. PMID 25573112
- [Background] Hirve S, Bavdekar A, Juvekar S, Benn CS, Nielsen J, Aaby P. Non-specific and sex-differential effects of vaccinations on child survival in rural western India. Vaccine. 2012 Nov 26;30(50):7300-8. doi: 10.1016/j.vaccine.2012.09.035. Epub 2012 Sep 26. PMID 23022401
- [Background] Aaby P, Andersen A, Ravn H, Zaman K. Co-administration of BCG and Diphtheria-tetanus-pertussis (DTP) Vaccinations May Reduce Infant Mortality More Than the WHO-schedule of BCG First and Then DTP. A Re-analysis of Demographic Surveillance Data From Rural Bangladesh. EBioMedicine. 2017 Aug;22:173-180. doi: 10.1016/j.ebiom.2017.07.012. Epub 2017 Jul 14. PMID 28784413
- [Background] Biering-Sorensen S, Aaby P, Lund N, Monteiro I, Jensen KJ, Eriksen HB, Schaltz-Buchholzer F, Jorgensen ASP, Rodrigues A, Fisker AB, Benn CS. Early BCG-Denmark and Neonatal Mortality Among Infants Weighing <2500 g: A Randomized Controlled Trial. Clin Infect Dis. 2017 Oct 1;65(7):1183-1190. doi: 10.1093/cid/cix525. PMID 29579158
- [Background] Higgins JP, Soares-Weiser K, Lopez-Lopez JA, Kakourou A, Chaplin K, Christensen H, Martin NK, Sterne JA, Reingold AL. Association of BCG, DTP, and measles containing vaccines with childhood mortality: systematic review. BMJ. 2016 Oct 13;355:i5170. doi: 10.1136/bmj.i5170. PMID 27737834
- See also: Related Info — https://www.bandim.org